CLINICAL TRIAL: NCT02399852
Title: Effects of Lomitapide on Carotid and Aortic Atherosclerosis in Patients Treated With Lomitapide in Usual Care (CAPTURE)
Brief Title: Effects of Lomitapide on Carotid and Aortic Atherosclerosis
Status: Withdrawn | Type: Observational
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AEGR-733-028
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2015-03

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lomitapide
  Other Names: Juxtapid; Lojuxta

SUMMARY:
Study to assess changes in carotid and aortic atherosclerosis in patients being treated with lomitapide.

DETAILED DESCRIPTION:
This is a multi-center long-term open-label non-comparative study to assess changes in carotid and aortic atherosclerosis in patients being treated with lomitapide. Patients from countries in the EU, the US and Canada who are being treated with lomitapide and are enrolled in The Lomitapide Observational Worldwide Evaluation Registry (LOWER), will be invited by the LOWER enrolling physician to participate in this substudy.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients (age ≥18 years) who are enrolled in LOWER

Exclusion Criteria:

* Patients with a prior history of carotid angioplasty, carotid stenting, or carotid atherectomy
* Patients with a contraindication to MRI examination (i.e., brain aneurysm, implanted neural stimulator, implanted cardiac pacemaker, pacemaker wires or defibrillator, prosthetic heart valves, cochlear implant, ocular foreign body, or other implanted body)
* Patients who have undergone a coronary stenting procedure in the preceding three weeks prior to enrollment
* Patients prone to claustrophobia or known anxiety disorders that will interfere with the ability to acquire quality MRI scans
* Patients with an implanted insulin pump
* Patients with metal shrapnel or bullet wounds
* Patients with a body mass index (BMI) > 40 kg/m2 (since it may be difficult to position comfortably with the MRI scanner)
* Patients who work with metal lathes (unless an orbit x-ray performed prior to the enrollment MRI scan has been done to rule out metal fragments in the eye)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in LOWER
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The percent change from baseline in cartoid vessel wall area at the two-year evaluation | 2 years

SECONDARY OUTCOMES:
The percent change from baseline to one and five years on therapy for carotid and aortic vessel wall area, and carotid and aortic vessel wall thickness. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Qing Chang, MD, Principal Investigator — Aegerion Pharmaceuticals, Inc.